CLINICAL TRIAL: NCT07336719
Title: The Effect of Showing Cartoons and Playing Music During Dental Treatment on Pain and Treatment Anxiety in Children: A Randomized Controlled Trial
Brief Title: The Effect of Cartoon and Music Applications on Dental Pain
Acronym: Pain Relief
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Sibel Küçükoğlu, Prof., Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 02-SU.01-2026SA/2025
Record Dates: First submitted 2026-01-02; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Pain Management; Dental Anxiety; Distraction; Dental Extraction
Keywords: anxiety; distraction; dental extraction; pain management; nursing care
MeSH Terms: conditions — Agnosia; Anxiety Disorders | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The G*Power 3.1.9.2 program was used to calculate the sample size for the study. The G*Power 3.1.9.6 program was used for the prior sample size calculation. Anticipating potential losses, the sample size was increased by approximately 20%, and the study was planned to be conducted with 20 children in each group.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimantal Group: Cartoon Group (Experimental): In this group of 20 children, cartoons were shown during the tooth extraction procedure. Before the procedure began, the child's vital signs (heart rate and blood oxygen level), pain level, and fear level were measured. The child watched their chosen cartoon during the procedure. Vital signs and pain level were measured again during the procedure. One minute after the procedure was completed, the child's vital signs, pain level, and fear level were measured again.
  Interventions: Other: Cartoon viewing app
- Experimantal Group: Music Group (Experimental): In this group of 20 children, music was played during the tooth extraction procedure. Before the procedure began, the child's vital signs (heart rate and blood oxygen level), pain level, and fear level were measured. The music chosen by the child was played during the procedure. Vital signs and pain level were measured again during the procedure, and again 1 minute after the procedure was completed.
  Interventions: Other: Music intervention
- Control Group (Other): The control group consisted of 20 children who underwent the routine procedure. One minute before the procedure, the child's vital signs (heart rate and blood oxygen level), pain level, and fear level were measured. Vital signs and pain level were measured again during the procedure. One minute after the procedure was completed, the child's vital signs, pain level, and fear level were measured again.
  Interventions: Other: control group

INTERVENTIONS:
Other: Cartoon viewing app — Before starting the study, a compilation of children's favorite cartoons specific to their age group was prepared. Based on randomization, children in this group were asked before the procedure which cartoon they would like to watch. During the procedure, a tablet was placed in a position where the child could easily see it. The cartoon started being shown one minute before the procedure. Uninterrupted viewing was ensured throughout the procedure.
  Arms: Experimantal Group: Cartoon Group
Other: Music intervention — Before starting the study, a list of children's favorite music specific to their age group was compiled. Children in this group were randomly assigned to listen to which music from this list before the procedure. Wireless headphones were placed on the child before the procedure. Music began playing one minute prior to the procedure. The child was allowed to listen to music continuously throughout the procedure.
  Arms: Experimantal Group: Music Group
Other: control group — No interventions were performed on the children in this group outside of routine practice.
  Arms: Control Group

SUMMARY:
This study investigated the effect of showing cartoons or playing music during the procedure on the physiological parameters of pain and fear experienced by children aged 6-12 undergoing tooth extraction treatment.

DETAILED DESCRIPTION:
Pediatric patients are frequently exposed to medical procedures that can cause pain and anxiety. While pharmacological interventions may be used, distraction is a simple and effective technique that diverts children's attention away from distressing stimuli. Distraction is a non-pharmacological pain management technique widely used by healthcare professionals during procedures to reduce pain and distress. It is based on the assumption that by shifting the child's attention to something interesting, their ability to pay attention to painful stimuli is inhibited, thereby reducing pain, distress, and anxiety. However, there are no published studies examining the effect of watching cartoons, listening to music, and the tell-show-do approach during tooth extraction on the physiological parameters, pain, and anxiety of children aged 6-12 years.

ELIGIBILITY:
Inclusion Criteria:

* Be between 6 and 12 years of age,
* Have no systemic, neurological, or chronic diseases,
* Agree to sit in the patient chair (according to the Frankl scale: 2, 3, or 4),
* Have no mental or neurological problems,
* Understand and speak Turkish,
* Have an indication for tooth extraction
* Willingness to participate in the study,
* No visual or auditory impairments

Exclusion Criteria:

* Being a foreign national,
* Not wanting to participate in the study,
* Not agreeing to sit in the patient chair (1 on the Frankl scale)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Child Identification Information Form | Five minutes before the procedure
  This form was created by researchers based on the literature to determine the identifying characteristics (age, gender, type and duration of treatment, etc.) of a child undergoing dental treatment.
Physiological Parameter Follow-up Form (Heart rate-min) | Tooth extraction 1 minute ago
  This is a form developed by researchers to assess the pulse and oxygen saturation of a child undergoing treatment.
Physiological Parameter Follow-up Form (oxygen saturation -SpO2%) | Tooth extraction 1 minute ago
  This is a form developed by researchers to assess the pulse and oxygen saturation of a child undergoing treatment.
Wong Baker Facial Pain Rating Scale | Tooth extraction 1 minute ago
  The Wong Baker Facial Rating Scale is one of the scales used to assess pain. This scale consists of six facial expressions, rated from 0 to 10 according to the severity of the pain.
Child Fear Assessment Scale-Dental Subscale (CFSS-DS) | Tooth extraction 1 minute ago
  The CFSS-DS scale consists of 15 questions covering different aspects of dental treatment. It can be used with children aged 4-14 years. It is used to determine children's fear of tooth extraction.

SECONDARY OUTCOMES:
Physiological Parameter Follow-up Form (Heart rate-min | 5th minute of the process
  This is a form developed by researchers to assess the pulse and oxygen saturation of a child undergoing treatment.
Physiological Parameter Follow-up Form (oxygen saturation -SpO2%) | 5th minute of the process
  This is a form developed by researchers to assess the pulse and oxygen saturation of a child undergoing treatment.
Wong Baker Facial Pain Rating Scale | 5th minute of the process
  The Wong Baker Facial Rating Scale is one of the scales used to assess pain. This scale consists of six facial expressions, rated from 0 to 10 according to the severity of the pain.
Physiological Parameter Follow-up Form (Heart rate-min) | 1 minute after the procedure
  This is a form developed by researchers to assess the pulse and oxygen saturation of a child undergoing treatment.
Physiological Parameter Follow-up Form (oxygen saturation -SpO2%) | 1 minute after the procedure
  This is a form developed by researchers to assess the pulse and oxygen saturation of a child undergoing treatment.
Wong Baker Facial Pain Rating Scale | 1 minute after the procedure
  The Wong Baker Facial Rating Scale is one of the scales used to assess pain. This scale consists of six facial expressions, rated from 0 to 10 according to the severity of the pain.
Child Fear Assessment Scale-Dental Subscale (CFSS-DS) | 1 minute after the procedure
  The CFSS-DS scale consists of 15 questions covering different aspects of dental treatment. It can be used with children aged 4-14 years. It is used to determine a child's fear of tooth extraction.

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Kucukoglu, Study Director — Selcuk University
Locations (1):
- Selcuk University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Koller D, Goldman RD. Distraction techniques for children undergoing procedures: a critical review of pediatric research. J Pediatr Nurs. 2012 Dec;27(6):652-81. doi: 10.1016/j.pedn.2011.08.001. Epub 2011 Oct 13. PMID 21925588